CLINICAL TRIAL: NCT01054898
Title: A RCT to Test the Effectiveness of a Telephone Intervention to Improve the Mental Health of Community Dwelling Women Abused by Their Intimate Partners
Brief Title: Effectiveness of a Telephone Intervention to Improve the Mental Health of Abused Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Agnes Tiwari, Professor and Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW 06-105 T/1130
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Battered Women
Keywords: depression; spouse abuse; intervention studies
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- advocacy intervention (Experimental): A 12-week telephone social support and empowerment intervention consisting of empowerment training, scheduled weekly telephone calls, and 24-hour access to a hotline for abused women
  Interventions: Behavioral: advocacy intervention
- Usual community services (Active Comparator): Standard care for abused women in the community
  Interventions: Behavioral: usual community services

INTERVENTIONS:
Behavioral: advocacy intervention — A 12-week telephone social support and empowerment intervention consisting of empowerment training, scheduled weekly telephone calls, and 24-hour access to a hotline for abused women
  Arms: advocacy intervention
Behavioral: usual community services — standard care for abused women in the community
  Arms: Usual community services

SUMMARY:
The purpose of this study is to determine if a telephone social support and empowerment intervention is more effective than usual community services in improving the mental health of community-dwelling women abused by their intimate partners.

DETAILED DESCRIPTION:
Depression is one of the most common mental health sequelae of intimate partner violence (IPV). Although a range of interventions have been tried to improve the mental health of women survivors of IPV, the results are inconclusive. In this trial, a 12-week advocacy intervention consisting of empowerment and telephone social support is provided to abused Chinese women in a community setting. Usual community services provide the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Chinese women 18 years of age or older
* Self-report of psychological, physical or sexual abuse by their current or former intimate partner in the previous 12 months
* Live or work in a community within the catchment area of a community centre designated for the proposed study

Exclusion Criteria:

* Perpetrator is not an intimate partner

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
depression | On completion of intervention and six months post-intervention

SECONDARY OUTCOMES:
perceived social support | On completion of intervention and six months post-intervention
health-related quality of life | On completion of intervention and six months post-intervention
intimate partner violence | On completion of intervention and six months post-intervention
safety behaviors | On completion of intervention and six months post-intervention
utilization of health services | On completion of intervention and six months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Tiwari, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong Kong SKH Lady MacLehose Centre, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Tiwari A, Fong DY, Wong JY, Yuen KH, Yuk H, Pang P, Humphreys J, Bullock L. Safety-promoting behaviors of community-dwelling abused Chinese women after an advocacy intervention: a randomized controlled trial. Int J Nurs Stud. 2012 Jun;49(6):645-55. doi: 10.1016/j.ijnurstu.2011.12.005. Epub 2012 Jan 9. PMID 22227168
- [Derived] Tiwari A, Fong DY, Yuen KH, Yuk H, Pang P, Humphreys J, Bullock L. Effect of an advocacy intervention on mental health in Chinese women survivors of intimate partner violence: a randomized controlled trial. JAMA. 2010 Aug 4;304(5):536-43. doi: 10.1001/jama.2010.1052. PMID 20682933